CLINICAL TRIAL: NCT00255268
Title: Longitudinal, Randomized, Open and Prospective Clinical Trial to Evaluate the Efficacy of Continuous vs Intermittent Maximum Androgen Blockade (CMAB vs IMAB) With Goserelin-Bicalutamide Combination in the Treatment of Hormonal naïve With Metastatic Prostate Cancer
Brief Title: CMAB vs IMAB in Metastatic Prostate Cancer
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D6876L00010
Record Dates: First submitted 2005-10-26; First posted 2005-11-18 (Estimated); Last update posted 2007-08-28 (Estimated); Status verified 2007-08

CONDITIONS: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Goserelin; bicalutamide

INTERVENTIONS:
Drug: Goserelin
Drug: Bicalutamide

SUMMARY:
To evaluate the efficacy, safety and survival of two treatment regimens: Continuous Intermittent Maximum Androgen Blockade, using goserelin and bicalutamide in patients with prostate cancer. Primary endpoint is time to progression. Fifteen patients will be evaluated. QoL evaluation is also included.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of D2 of Adenocarcinoma,
* Naivety to treatment
* Valuable bone metastasis

Exclusion Criteria:

* Hematological, liver or renal toxicity Grade IV
* Severe and active infections

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2004-08

PRIMARY OUTCOMES:
Time to progression

SECONDARY OUTCOMES:
Safety
Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Mexico Medical Director, MD, Study Director — AstraZeneca
Locations (2):
- Mexico (2):
  - Research Site, Metepec
  - Research Site, Mexico City